CLINICAL TRIAL: NCT05042557
Title: Real World Study of Diagnosis, Treatment and Prognosis of Malignant Pleural Mesothelioma in China
Brief Title: Real World Study of MPM in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zhouguang Hui, M.D., M.D., Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: NCC202062402
Record Dates: First submitted 2021-09-05; First posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Malignant Pleural Mesothelioma; Diagnoses Disease; Treatments; Prognosis
Keywords: MPM; Prognosis; Radiotherapy
MeSH Terms: conditions — Mesothelioma, Malignant

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Sun Yat-sen University Cancer Center
- hanghai Chest Hospital
- Tianjin Cancer Hospital
- Fudan University Shanghai Cancer Center
- Anhui Cancer Hospital
- Shandong Cancer Hospital
- Hunan Cancer Hospital
- Yunnan Cancer Hospital
- Chinese Academy of Medical Sciences

SUMMARY:
Malignant pleural mesothelioma (MPM) is a highly aggressive tumor with atypical clinical manifestations. Most patients with MPM are at an advanced stage at the time of diagnosis, and only a few patients can be cured by radical surgery and other treatment measures. Pemetrexed + cisplatin chemotherapy with or without bevacizumab is still the standard treatment for MPM. In recent years, multimodality therapy including surgery, radiotherapy and chemotherapy have shown certain advantages in improving patient overall survival time. Targeted and immunotherapy may bring breakthroughs in MPM therapy. However, there are still no high-quality evidence-based medical evidence reports on the treatment model and effects of MPM patients in China.

Focusing on MPM, we plan to systematically review the relevant scientific literature, confirm relevant scientific research questions, and provide references for related treatments. On this basis, we will estimate MPM incidence and mortality rates from 2014 to 2025 based on the data published by the National Cancer Registry. Meanwhile, a retrospective study cohort was constructed based on the electronic medical record database, and according to the research demand, patients were followed up with their post-discharge survival status to comprehensively describe and analyze the incidence, diagnosis, treatment, and prognosis of MPM patients. Also, exploratory analysis of the therapeutic effects of existing clinical treatments was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed as malignant pleural mesothelioma
* Aged over 18

Exclusion Criteria:

* Follow-up less than 3 months

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who were pathologically confirmed as malignant pleural mesothelioma is included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2-year overall survival
  Overall survival is defined as the time from diagnosis to death for any reason or last follow-up

SECONDARY OUTCOMES:
Progression-free survival | 2-year progression-free survival
  Progression-free survival is defined as the time from diagnosis to the first event of progression

CONTACTS AND LOCATIONS:
Overall Officials: Zhouguang Hui, Ph.D., Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China